CLINICAL TRIAL: NCT02442336
Title: A Web-based Multimedia Intervention for Head and Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB11822
Record Dates: First submitted 2015-03-18; First posted 2015-05-13 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: Cancer of the Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- My Journey AHead (Experimental): Several internet modules will be developed to address mouth and swallowing concerns, oral care, healthy eating, speech problems, coping with cancer, pain management, and physical therapy.
  Interventions: Behavioral: My Journey AHead

INTERVENTIONS:
Behavioral: My Journey AHead — The intervention program will contain information and interactive activities around swallowing concerns, proper oral care, healthy eating and nutrition, speech issues, stress and coping with cancer, and pain management.

SUMMARY:
The overall goal is to develop and examine the acceptability of a web-based (Internet) intervention program for patients with head and neck cancer who have recently completed radiation therapy.

DETAILED DESCRIPTION:
The overall goal is to develop and examine the acceptability of a theory-guided, web-based multimedia intervention program for head and neck cancer patients who have recently completed radiation therapy. The effects of this intervention on patients' quality of life (QOL) will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx
* Are receiving or have completed radiation therapy within in the past 12 months

Exclusion Criteria:

* Inability to read and/or communicate in English
* Head and neck cancers of non-squamous histology (e.g., adenoid cystic carcinoma, adenocarcinoma, sarcoma)
* Blindness or severity of visual impairment that precludes one's ability to view images/text
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-06-15 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Fang, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Fang CY, Longacre ML, Manne SL, Ridge JA, Lango MN, Burtness BA. Informational Needs of Head and Neck Cancer Patients. Health Technol (Berl). 2012 Apr 1;2(1):57-62. doi: 10.1007/s12553-012-0020-9. Epub 2012 Feb 14. PMID 22518350
- [Derived] Fang CY, Galloway TJ, Egleston BL, Bauman JR, Ebersole B, Chwistek M, Buhler JG, Longacre ML, Ridge JA, Manne SL, Manning C. Development of a Web-Based Supportive Care Program for Patients With Head and Neck Cancer. Front Oncol. 2020 Dec 15;10:602202. doi: 10.3389/fonc.2020.602202. eCollection 2020. PMID 33384959

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | My Journey AHead
Started | 80
Developmental Phase | 6
Evaluation Phase | 74
Provided Access to Intervention (55 participants were provided access to My Journey AHead. 44 participants logged in and viewed the program, whereas 11 participants did not log in or access the program.) | 55
Completed | 44
Not Completed | 36
Not completed — 6 patients assisted with the intervention development only. | 6
Not completed — Of the 74 who consented, 19 did not complete baseline assessment and were withdrawn from the study. | 19
Not completed — Lost to Follow-up | 11

BASELINE CHARACTERISTICS:
Groups:
- My Journey AHead: Participants were provided access to a web-base intervention that included several modules on oral care, stress and coping, nutrition, and pain management.
Arm/Group | My Journey AHead
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.1 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 49
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 55
Brief Symptom Inventory-18 [Mean (Standard Deviation); unit: units on a scale] — The Brief Symptom Inventory-18 (BSI-18) is an 18-item instrument widely used to measure psychological distress. The BSI-18 yields a total score (Global Severity Index), which is a measure of overall psychological distress. Raw scores are converted to t-scores (range 0-100) based on gender-specific normative data from cancer patient populations. A t-score of 50 is equal to the mean of the population. Higher scores represent greater levels of distress.
  units on a scale | 67.04 (4.123)
Cancer Behavior Inventory (CBI-B) [Mean (Standard Deviation); unit: units on a scale] — Self-efficacy for coping with cancer-related stressors and activities was assessed using the brief version of the Cancer Behavior Inventory (CBI-B), which at the time was a 14-item shortened version of the original CBI. The CBI-B is intended to be a single score measure of coping self-efficacy. Response options range from 1 to 9, and scores are summed across all items to create a total score (range = 14-126). Higher scores indicate greater coping efficacy.
  units on a scale | 92.25 (12.70)

OUTCOME MEASURES:

1. Primary Outcome: Patient Distress
Description: Psychological distress will be assessed using the Brief Symptom Inventory-18. The Brief Symptom Inventory-18 (BSI-18) is an 18-item scale widely used to measure psychological distress. The BSI-18 yields a total score (Global Severity Index), which is a measure of overall psychological distress. Raw scores are converted to t-scores (range 0-100) based on gender-specific normative data from cancer patient populations. A t-score of 50 is equal to the mean of the population. Higher scores represent greater levels of distress. The BSI-18 provides a clinical case-rule classifying respondents who have a t-score score ≥ 63 on the GSI as having clinically significant symptoms. Other studies have used a lower cutoff, with a GSI t-score ≥ 57 recommended as a cutoff for clinically significant symptoms in a study of cancer patients.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Web-Based Intervention: Participants were provided access to a web-base intervention that included several modules on oral care, stress and coping, nutrition, and pain management.
Arm/Group | Web-Based Intervention
Number analyzed (Participants) | 44
units on a scale | 66.16 (4.77)

ADVERSE EVENTS:
Time Frame: A 3- to 6-week period during which participants were on-study (i.e. consented, completed baseline assessment, provided access to the intervention, and completed program evaluation).
Description: Adverse events due to clinical treatment or medical management of the patient's disease were not specifically collected in this behavioral study, unless the patient reported it to the study team. We did not obtain IRB approval to conduct a medical chart review for incidence of treatment-related adverse events.
Arm/Group | My Journey AHead
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 50/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | My Journey AHead (N=55)
Elevated distress (Psychiatric disorders) | 50 (50) — High levels of psychological distress (above the established cutoff score of >= 63 on the BSI-18) were reported at baseline by 50 of the 55 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT02442336/Prot_SAP_000.pdf